CLINICAL TRIAL: NCT02399397
Title: Influence of Sepsis, Age and SLCO1A2 Genetic Polymorphisms on Rocuronium Pharmacokinetics-pharmacodynamics in ASA I-III Surgical Patients
Brief Title: Influence of Age, Sepsis and SLCO1A2 Polymorphisms on Rocuronium Pharmacokinetics
Acronym: ROCSEPSIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Natalia Valadares de Moraes, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROC1314730-0
Record Dates: First submitted 2015-03-02; First posted 2015-03-26 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-10

CONDITIONS: Sepsis; Systemic Inflammatory Response Syndrome; Septic Shock
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome; Shock, Septic | interventions — Hematologic Tests; Liver Extracts; Anesthesia, General; Midazolam; Rocuronium; Fentanyl; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Active Comparator): Adult patients(18-50 years old) ASA I-II without sepsis submitted to small to medium sized surgery under general anesthesia are being recruited. All patients are being induced with individualized doses of rocuronium, midazolam, propofol and fentanyl. Serial blood sampling are being collected up to 6 h after administration of the drug for pharmacokinetic study. Neuromuscular blockade is being monitored by stimulation of the adductor muscle of the thumb on the ulnar nerve through the train of four monitoring (TOF) at the same time as blood sampling. All patients are being submitted to blood testing for liver and renal function (creatinine, urea, albumin, aspartate aminotransferase and alanine aminotransferase).
  Interventions: Procedure: Serial blood sampling; Procedure: Train of four monitoring; Procedure: Blood testing for liver and renal function; Drug: General anesthesia; Procedure: Small to medium sized surgery under general anesthesia
- Sepsis group (Experimental): Adult patients (18-50 years old) ASAII and III with sepsis, systemic inflammatory response syndrome or septic shock submitted to small to medium sized surgery under general anesthesia are being recruited. All patients are being induced with individualized doses of rocuronium, midazolam, propofol and fentanyl. Serial blood sampling are being collected up to 6 h after administration of the drug for pharmacokinetic study. Neuromuscular blockade is being monitored by stimulation of the adductor muscle of the thumb on the ulnar nerve through the train of four monitoring (TOF) at the same time as blood sampling. All patients are being submitted to blood testing for liver and renal function (creatinine, urea, albumin, aspartate aminotransferase and alanine aminotransferase).
  Interventions: Procedure: Serial blood sampling; Procedure: Train of four monitoring; Procedure: Blood testing for liver and renal function; Drug: General anesthesia; Procedure: Small to medium sized surgery under general anesthesia
- Elderly group (Experimental): Elderly patients (> 65 years old) ASA I-II without sepsis submitted to small to medium sized surgery under general anesthesia are being recruited. All patients are being induced with individualized doses of rocuronium, midazolam, propofol and fentanyl. Serial blood sampling are being collected up to 6 h after administration of the drug for pharmacokinetic study. Neuromuscular blockade is being monitored by stimulation of the adductor muscle of the thumb on the ulnar nerve through the train of four monitoring (TOF) at the same time as blood sampling. All patients are being submitted to blood testing for liver and renal function (creatinine, urea, albumin, aspartate aminotransferase and alanine aminotransferase).
  Interventions: Procedure: Serial blood sampling; Procedure: Train of four monitoring; Procedure: Blood testing for liver and renal function; Drug: General anesthesia; Procedure: Small to medium sized surgery under general anesthesia

INTERVENTIONS:
Procedure: Serial blood sampling — Serial blood samples are being collected at times 0, 2, 5, 10, 15, 20, 30, 60, 120, 180, 240 and 360 minutes after rocuronium administration.
Procedure: Train of four monitoring — Neuromuscular blockade is being evaluated at the same time of blood sampling by stimulation of the adductor muscle of the thumb on the ulnar nerve through the train of four monitoring (TOF).
  Other Names: TOF
Procedure: Blood testing for liver and renal function — Blood testing: urea, creatinine, aspartate aminotransferase, alanine aminotransferase, albumin, glycemia
Drug: General anesthesia — All patients were induced with individual intravenous doses of midazolam, rocuronium, fentanyl and propofol.
  Other Names: Midazolam; Rocuronium; Fentanyl; Propofol
Procedure: Small to medium sized surgery under general anesthesia — Patients classified according American Society of Anesthesiologists (ASA) as ASA I-III and submitted to small-medium sized surgery under general anesthesia were recruited for the present investigation.

SUMMARY:
This study aims to evaluate the influence of age and sepsis on in vivo activity of OATP1A2 using rocuronium (ROC) as a probe and evaluating the pharmacokinetics and pharmacodynamics in ASA I-III surgical patients. Thus, adult patients without sepsis (control group, n= 12), adult patients with sepsis (sepsis group, n= 12) and elderly patients without sepsis (elderly group, n= 12), all submitted to small to medium-sized surgeries who were induced with individual doses of rocuronium, fentanyl and propofol are being investigated.

DETAILED DESCRIPTION:
Rocuronium (ROC), a neuromuscular blocking agent used in surgical procedures, is primarily eliminated by biliary excretion. Its distribution to the liver, mediated the organic anion transporting polypeptide 1A2 (OATP1A2), is a determining factor for the duration of neuromuscular blockade. Age and release of cytokines during inflammation and infection processes of sepsis can alter expression of SLCO1A2 gene, encoding OATP1A2. The objective of this study is to evaluate the influence of age and sepsis on in vivo activity of OATP1A2 using ROC as a probe and evaluating the pharmacokinetics and pharmacodynamics in ASA I-III surgical patients. Adult patients without sepsis (control group, n=12), adult patients with sepsis (sepsis group, n=12) and elderly patients without sepsis (elderly group, n=12), all submitted to small to medium-sized surgeries are being investigated. All patients are being induced with individual doses of rocuronium, fentanyl and propofol. Serial blood samples are being collected up to 360 minutes after administration of ROC. Neuromuscular blockade induced by ROC is monitored by stimulation of the adductor muscle of the thumb on the ulnar nerve through the train of four monitoring (TOF) at the same times of blood sampling. The plasma concentration of ROC will be analyzed by liquid chromatography coupled to mass spectrometry with electrospray ionization using positive ion mode.

ELIGIBILITY:
Inclusion Criteria:

* Adult and elderly patients, both gender.
* Patients submitted to small to medium-sized surgeries.
* Patients who were induced with individual doses of rocuronium, fentanyl and propofol.
* Patients with normal renal function (creatinine clearance > 60 mL/min).
* Patients with normal liver function.

Exclusion Criteria:

* Patients who were in use of fluoxetine, carbamazepine, aminoglycoside antibiotics, OATP1A2 inhibitors.
* Patients with gastrointestinal and liver diseases, neuromuscular disorders.
* Patients who were in chronic use of drugs which alter rocuronium effect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determination of AUC/dose | Up to 6h after rocuronium administration
  Determination of area under the plasma concentration versus time curve (AUC)/dose of rocuronium will be estimated for pharmacokinetic analysis.

SECONDARY OUTCOMES:
Determination of total clearance | Up to 6h after rocuronium administration
  Determination of total clearance of rocuronium will be estimated for pharmacokinetic analysis.
Determination of volume of distribution | Up to 6h after rocuronium administration
  Determination of volume of distribution of rocuronium will be estimated for pharmacokinetic analysis.
Determination of mean residence time | Up to 6h after rocuronium administration
  Determination of mean residence time of rocuronium will be estimated for pharmacokinetic analysis.
OATP1A2 genotyping using Real Time-PCR | Up to 5 minutes before rocuronium administration
  The single nucleotide polymorphisms of SLCO1A2 gene (404A>T, 559G>A, 833delA at coding sequence and -1105G>A, -1032G>A, -715T>C, -361G>A e -189_-188insA at the non-coding sequence of SLCO1A2) are being evaluated in all included patients, using Real Time PCR.
Analysis of cytokine IL-1α in plasma | Up to 5 minutes before rocuronium administration; 30 and 360 minutes after rocuronium administration
  Plasma cytokine Interleukin-1α (IL-1α) will be evaluated in each patient.
Analysis of cytokine IL-1β in plasma | Up to 5 minutes before rocuronium administration; 30 and 360 minutes after rocuronium administration
  Plasma cytokine IL-1β will be evaluated in each patient.
Analysis of cytokine IL-6 in plasma | Up to 5 minutes before rocuronium administration; 30 and 360 minutes after rocuronium administration
  Plasma cytokine IL-6 will be evaluated in each patient.
Analysis of cytokine TNF-α in plasma | Up to 5 minutes before rocuronium administration; 30 and 360 minutes after rocuronium administration
  Plasma cytokine Tumor Necrosis Factor-α (TNF-α) will be evaluated in each patient.
Pharmacokinetic-Pharmacodynamic analysis: relationship between rocuronium plasma concentration and the neuromuscular blockade | Up to 6h after rocuronium administration
  The relationship between rocuronium plasma concentration and the neuromuscular blockade will be described by a sigmoid maximum effect model for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Natalia V. de Moraes, Prof., Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, Araraquara, São Paulo, Brazil

REFERENCES:
- [Result] de Moraes NV, Lauretti GR, Filgueira GC, Lopes BC, Lanchote VL. Analysis of rocuronium in human plasma by liquid chromatography-tandem mass spectrometry with application in clinical pharmacokinetics. J Pharm Biomed Anal. 2014 Mar;90:180-5. doi: 10.1016/j.jpba.2013.11.032. Epub 2013 Dec 7. PMID 24370612
- [Derived] Costa ACC, Coelho EB, Lanchote VL, Correia BV, Abumansur JT, Lauretti GR, de Moraes NV. The SLCO1A2 -189_-188InsA polymorphism reduces clearance of rocuronium in patients submitted to elective surgeries. Eur J Clin Pharmacol. 2017 Aug;73(8):957-963. doi: 10.1007/s00228-017-2243-1. Epub 2017 Apr 14. PMID 28409297